CLINICAL TRIAL: NCT00278733
Title: Campus Health Intervention Projects to Reduce High Risk Drinking Among University Students by Means of Brief Physician Advice
Brief Title: Campus Health Intervention Projects UBC Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: B05 0636
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: High Risk Drinking
Keywords: Randomized controlled trial; brief intervention; university students; physician advice; high risk drinking
MeSH Terms: interventions — Crisis Intervention

INTERVENTIONS:
Behavioral: Brief intervention (physician advice)

SUMMARY:
The goal of the study is to test the efficacy of brief physician advice in reducing the frequency of high risk drinking and alcohol-related harm in a population of university students seeking routine care at UBC Student Health Service. It is hypothesized that receiving the intervention will reduce the amount of alcohol consumed and the incidence of alcohol-related harm among the students in the intervention group, as compared to the control group.

DETAILED DESCRIPTION:
We estimate that roughly 3000 students will need to be screened to obtain sufficient eligible participants to randomize 150 students. High-risk drinkers will be identified by means of an embedded alcohol screening survey, which will be distributed through Student Health Services. Those deemed eligible through the screening survey and who have agreed to be contacted will be invited to attend a baseline interview, which will further define eligibility and assign interested students to the control or intervention group. Those randomized to the usual care control group will receive a self-help health booklet and will be contacted to complete a follow-up telephone interview at 6, 12, 18 and 24 months. Those randomized to the intervention group will receive the same booklet and will meet with a Student Health Service physician. There will be two face-to-face meetings with the physician and two follow up phone calls by the physician. The physicians use a scripted workbook, diary cards and other materials designed to reduce alcohol use and the frequency of high risk drinking. Those in the intervention group will also be contacted to complete a follow-up telephone interview at 6, 12, 18 and 24 months. Outcome data will also be sought, with participants' permission, from campus organizations including Campus Housing, Security, the RCMP and the Registrar.

ELIGIBILITY:
Inclusion Criteria:

Full time students 18 and older; students seeking routine care at UBC Student Health Services; students who report high risk drinking in the last 28 days; students able to read and communicate in English

Exclusion Criteria:

Students graduating or leaving campus before the first intervention is complete; students who are acutely ill; students who are under 18 years; female students who are pregnant; students who are suicidal; students consuming more than 200 drinks in the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-02; Study Completion 2008-05

PRIMARY OUTCOMES:
A reduction in alcohol use and in the frequency of high risk drinking and related harms, measured at 6, 12, 18 and 24 months post intervention.

SECONDARY OUTCOMES:
Academic performance; contact with Campus Security or RCMP; incidents reported by campus housing; hospitalizations for injury or accident, as measured at 6, 12 18 and 24 months post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Saewyc, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- UBC Student Health Service, Vancouver, British Columbia, Canada